CLINICAL TRIAL: NCT03404323
Title: "Retinal Thickness Change Following Cataract Surgery in Eyes With Epiretinal Membrane"
Brief Title: "Cataract Surgery in Eyes With Epiretinal Membrane"
Status: Completed | Type: Observational
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Barbara Wetzel, Principal Investigator, St John of God Hospital, Vienna
Other Study IDs: 15062015
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Epiretinal Membrane; Pseudophakic Cystoid Macular Edema; Irvine-Gass Syndrome; Cataract
Keywords: central retinal thickness; epiretinal membrane; cataract surgery; pseudophakic cystoid macular edema
MeSH Terms: conditions — Epiretinal Membrane; Macular Edema; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to evaluate retinal thickness change and the occurrence of central structural retinal changes after uneventful small-incision cataract surgery in eyes with asymptomatic early stages of epiretinal membrane.

DETAILED DESCRIPTION:
Optical coherence tomography (OCT) is nowadays used in daily clinical practice and has become a helpful tool for detection of macular changes also in presence of opacification of the lens before cataract surgery. Using recent high-resolution OCT technology, early stages of epiretinal membranes can easily be detected and analysed. Since cataract surgery is one of the most frequently performed operations worldwide, this study was aimed to investigate the influence of uncomplicated cataract surgery on central retinal thickness and the incidence of structural and morphological macular changes after surgery in eyes with asymptomatic epiretinal membrane.

ELIGIBILITY:
Inclusion Criteria:

* visually compromising cataract and asymptomatic early stages of epiretinal membrane with no structural changes such as cysts or photoreceptor distribution in optical coherence tomography.

Exclusion Criteria:

* visual impairment or metamorphopsia due to epiretinal membrane
* history of branch retinal vein occlusion
* central retinal vein occlusion
* wet or dry macular degeneration
* diabetic retinopathy
* uveitis or other inflammatory eye disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty patients with visually compromising cataract and asymptomatic epiretinal membrane (ERM group) and 15 consecutive eyes with senile cataract with a healthy macula (control group) were included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
central macular thickness | Change from Baseline central macular thickness at 3 months
  Central 1-millimeter and 3-milimeter retinal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Wetzel, MD, Principal Investigator — St John of God Hospital, Vienna; Georgios Mylonas, MD, Study Director — St John of God Hospital, Vienna